CLINICAL TRIAL: NCT06343298
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO-CONTROLLED, DOSE TITRATION, MULTI-CENTER STUDY TO EVALUATE THE SAFETY AND EFFICACY OF SUBCUTANEOUS MANP WHEN ADMINISTERED ONCE DAILY FOR 42 DAYS IN PARTICIPANTS WITH DIFFICULT TO CONTROL HYPERTENSION/RESISTANT HYPERTENSION
Brief Title: To Evaluate the Safety and Efficacy of MANP in Subjects With Difficult to Control/ Resistant Hypertension
Acronym: BOLD-HTN
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: E-Star BioTech, LLC (Industry)
Collaborators: Mayo Clinic (Other); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ES_MANP_2001
Record Dates: First submitted 2024-03-20; First posted 2024-04-02 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-03

CONDITIONS: Difficult to Control Hypertension
Keywords: Resistant Hypertension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo-matched control (Placebo Comparator): Placebo-matched vehicle (vehicle minus the active component)
  Interventions: Other: Placebo Matched control
- MANP (Active Comparator): MANP in vehicle
  Interventions: Drug: MANP

INTERVENTIONS:
Drug: MANP — MANP (modified atrial natriuretic peptide) is a peptide that is being developed for treatment of difficult to control/resistant hypertension.
  Arms: MANP
Other: Placebo Matched control — This is a placebo matched vehicle - Vehicle minus the active ingredient
  Arms: Placebo-matched control

SUMMARY:
This is a Phase 2 dose-titration study designed to evaluate the safety and efficacy of MANP subcutaneous injection compared to placebo in reducing baseline daytime systolic blood pressure (SBP), derived from 24-hour ambulatory blood pressure monitoring (ABPM), in subjects with hypertension who are taking 3 or more antihypertensive medications with different mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for enrollment in the study only if they meet ALL the following criteria at time of Screening:

* Male or female subjects aged 18 - 80 years, inclusive, at the screening visit.
* Female subjects must not be of childbearing potential
* Subjects must be taking appropriate doses of 3 or more antihypertensive drugs with different mechanisms of action. One of which must be a diuretic and the other must be an ACEi or ARB at atleast 50% of the maximum recommended dose for hypertension.
* Subjects must have a seated (5 minutes) systolic blood pressure ≥ 140 mmHg and SBP ≥135 mmHg by ABPM prior to randomization (T1).
* Subjects must have a CKD-EPI eGFR ≥ 30 mL/min/1.73m2
* A subset of the subjects with an eGFR between 20-30 ml/min/1.73m2 will be included, not to exceed 10% of the total study subjects.
* Subjects must have a BMI between 18 - 40 kg/m2.
* Subjects who engage in sexual intercourse in which their partner could become pregnant must agree to use a barrier method of birth control (i.e., vaginal/penile condom) with spermicide for the duration of the study and for 90 days after the last dose of study drug or be at least 6 weeks post-vasectomy with confirmation by post-vasectomy semen analysis. In addition, subjects may not donate sperm for the duration of the study and for 90 days after the last dose of study drug.

Exclusion Criteria:

Subjects meeting ANY of the following criteria at time of Screening will be excluded from enrollment:

* Subjects with an average sitting systolic blood pressure ≥180 mmHg or diastolic blood pressure ≥ 110 mmHg at Screening (SV), or prior to randomization at T1.
* Subjects with a history of secondary hypertension, including but not limited to coarctation of the aorta, primary hyperaldosteronism, renal artery stenosis, Cushing's disease, pheochromocytoma, and polycystic kidney disease. If the subject has not previously been evaluated for secondary hypertension, investigators are responsible for evaluating all potential secondary causes of hypertension in accordance with current practices and clinical guidelines before entering the patient into the study.
* Subjects with an HbA1c ≥ 8% at screening (SV)
* Subjects who have experienced myocardial infarction, unstable angina, or a cerebrovascular accident (CVA) within 6 months of the Screening Visit; or sick sinus syndrome or second- or third-degree atrioventricular block, or recurrent atrial tachyarrhythmia, recurrent ventricular tachycardia, or symptomatic bradycardia.
* Subjects who have an implanted cardioverter defibrillator (ICD) that has been fired for any arrhythmia within 3 months of Screening (SV) or implanted pacemakers.
* Subjects with congestive heart failure (New York Heart Association [NYHA] class II-IV)
* Subjects with hemodynamically significant valvular heart disease
* Subjects undergoing hemodialysis or peritoneal dialysis, or history of renal transplant.
* Subjects who have diagnosis or recurrence of malignancy within the past 3 years
* Subjects with a documented history of sleep apnea, with a prescription for CPAP therapy.
* Women of childbearing potential
* Subjects who are pregnant or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-17 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mean daytime SBP derived from 24-hour ABPM at approximately Day 42. | Approximately 42 days
  ABPM
Incidence and severity of Adverse events through 4- weeks post end of treatment. | Approximately 10 weeks
  Safety
Incidence and severity of Serious Adverse Events through 4- weeks post end of treatment. | Approximately 10 weeks
  Safety
Incidence and severity of Treatment Emergent Adverse Events through 4- weeks post end of treatment. | Approximately 10 weeks
  Safety

SECONDARY OUTCOMES:
Change in Clinic sitting systolic blood pressure | Approximately 42 days
  Achieving mean seated (5 minutes) systolic blood pressure blood pressure control ≤ 130 mmHg at end of treatment visit.
Pharmacokinetics - Cmax | Approximately 42 days
  Maximum concentration of MANP in plasma post dose on Day 1 and Last day of Treatment
Pharmacokinetics - Tmax | Approximately 42 Days
  Time required to achieve maximum concentration of MANP in plasma post dose on Day 1 and Last day of Treatment
Anti-drug Antibody | Approximately 10 weeks
  Change in Anti-drug antibodies against MANP and ANP at Days 21 and 42 post treatment and at follow up visits 1 and 2 compared to baseline

OTHER OUTCOMES:
Differential Outcomes in African-American Subject versus Non-African American Subjects | Approximately 42 days
  Change mean daytime SBP from ABPM, from baseline compared to end of treatment visit in African American population and the non-African American population at each dose level.
Metabolic biomarkers - Glucose | Approximately 10 weeks
  Change from baseline in plasma Glucose at end of treatment and Follow-up
Metabolic biomarkers - Insulin | Approximately 10 weeks
  Change from baseline in plasma Insulin at end of treatment and Follow-up
Metabolic biomarkers - HbA1C | Approximately 10 weeks
  Change from baseline in HbA1C at end of treatment and Follow-up
Lipid biomarkers - HDL | Approximately 10 weeks
  Change from baseline in plasma High density Lipoprotein (HDL) at end of treatment and Follow-up
Lipid biomarkers - LDL | Approximately 10 weeks
  Change from baseline in plasma Low density Lipoprotein (LDL) at end of treatment and Follow-up
Lipid biomarkers - TG | Approximately 10 weeks
  Change from baseline in plasma Triglycerides (TG) at end of treatment and Follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David Smith, MD, Study Director — E-Star BioTech, LLC
Locations (29):
- United States (29):
  - Lynn Institute of the Ozarks, Little Rock, Arkansas
  - Amicis Research Center - Beverly Hills, Beverly Hills, California
  - Amicis Research Center - Granada Hills, Granada Hills, California
  - Orange County Research Center, Lake Forest, California
  - Amicis Research Center - Palmdale, Palmdale, California
  - Amicis Research Site - Valencia, Valencia, California
  - Interventional Cardiology Medical Group, West Hills, California
  - Office of Dr. Edward Portnoy MD, Westlake Village, California
  - SM Research Center, Biscayne Park, Florida
  - Arrow Clinical Trials, Daytona Beach, Florida
  - Royal Research Corp, Hollywood, Florida
  - Evolution Clinical Trials, Miami, Florida
  - Cowry Health, Acworth, Georgia
  - Alta Pharmaceutical Research Center, Peachtree Corners, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Revival Research Institute, LLC, Dearborn, Michigan
  - Aa Mrc Llc, Flint, Michigan
  - Monroe Biomedical Research, Monroe, North Carolina
  - Superior Clinical Research, Smithfield, North Carolina
  - K&R Research LLC, Marion, Ohio
  - Tristar Clinical Investigations, P.C., Philadelphia, Pennsylvania
  - Prime Research, Coppell, Texas
  - Dallas Renal Group, Dallas, Texas
  - East Texas Cardiology, Houston, Texas
  - Pioneer Research Solutions, Houston, Texas
  - Prime Clinical Research, Mansfield, Texas
  - Clinical Investigations of Texas, Plano, Texas
  - Aavon Clinical Trials, Richmond, Texas
  - Revival Research, Sherman, Texas

IPD SHARING:
Plan to Share IPD: Yes
All IPD that support publications
Supporting Information: Study Protocol, CSR
Time Frame: As needed for publication support
Access Criteria: IPD will be shared with approved collaborators
URL: https://www.e-star.bio/